CLINICAL TRIAL: NCT07322302
Title: Repeat Eyelid Surgery for Trichiasis: Optimizing Results in East Africa (RESTORE): A Randomized Controlled Trial Comparing Two Surgical Techniques for Repeat Trichiasis Surgery Performed by Integrated Eye Care Workers
Brief Title: RESTORE: Comparing Two Approaches to Repeat TT Surgery Performed by Integrated Eye Care Workers (IECWs)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Virginia (Other); University of Pennsylvania (Other); Kongwa Trachoma Project (Unknown); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-2957; 1UG1EY036891 (NIH)
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Trachoma; Eye Diseases; Trichiasis
Keywords: Surgery; Oculoplastics; trichiasis; trachoma
MeSH Terms: conditions — Trachoma; Eye Diseases; Trichiasis

STUDY DESIGN:
Intervention Model Description: 1:1 randomization at the person level, stratified by surgeon and baseline PTT severity (mild vs severe)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and outcome examiners will be masked to treatment assignment. Field-based outcomes will be assessed in the field by masked outcome examiners (e.g. presence of rPTT, granuloma), and photograph-based outcomes (e.g., ECA) will be graded centrally at the data coordinating center in a masked fashion. Given the nature of the study, surgeons will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevel/rotate/advance procedure (B-RAP) (Experimental): Trichiasis surgery using the B-RAP procedure.
  Interventions: Procedure: B-RAP
- Bilamellar tarsal rotation (BLTR) (Active Comparator): Trichiasis surgery using the BLTR procedure.
  Interventions: Procedure: BLTR

INTERVENTIONS:
Procedure: B-RAP — B-RAP uses an incision beveled toward the eyelashes to thin the distal fragment and allow access to and removal of scarring from previous surgery. The distal fragment is rotated and the tarsus and conjunctiva are advanced downward to further correct the PTT.
  Arms: Bevel/rotate/advance procedure (B-RAP)
Procedure: BLTR — A full-thickness incision is made through the anterior and posterior lamellae, parallel to and 3mm above the lid margin. Three sutures are placed externally to rotate and fix the eyelid.
  Arms: Bilamellar tarsal rotation (BLTR)

SUMMARY:
The primary objective of this randomized clinical trial is to determine whether repeat trichiasis surgery performed with Bevel-Rotate Advancement Procedure (B-RAP) improves surgical success compared to Bilamellar Tarsal Rotation (BLTR) among a group of 8-10 TT surgeons in Tanzania. The study aims to enroll 1,000 individuals with PTT. The primary outcome is repeat PTT within one year after surgery. Additionally, the study will assess eyelid contour abnormalities and how they change over a two-year period as well as patient reported outcomes.

If this project is successful in improving surgical outcomes, it could change the approach to treating PTT globally. Individuals with trichiasis have a significantly reduced quality of life; correcting their trichiasis long-term has the potential to improve their quality of life and their family members' quality of life considerably.

DETAILED DESCRIPTION:
The investigators will randomize 1000 individuals with post-operative trichiasis on a 1:1 basis to standard BLTR surgery or the recently developed Bevel-Rotate Advancement Procedure (B-RAP). Participants will receive trichiasis surgery and will be followed at 1 day, 2 weeks and 3, 6, 9 12, 18 and 24 months after surgery. The primary outcome is development of repeat post-operative trachomatous trichiasis (rPTT) within 12 months after surgery. Logistic regression analyses will be performed to compare the rates of PTT between the two procedures, controlling for demographic characteristics and pre-operative trichiasis severity.

Secondary outcomes include pyogenic granuloma formation and eyelid contour abnormalities as well as patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* One or both eyes with upper eyelid PTT, with a plan to undergo PTT surgery
* Previous upper eyelid TT surgery in the study eye(s)
* Collection of all baseline data prior to randomization
* Signed, informed consent

Exclusion Criteria:

* Unable to provide informed consent
* All eyes with previously operated trichiasis that are phthisical

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of eyelids with repeat postoperative trachomatous trichiasis (rPTT) within 12 months after surgery | >2 weeks after surgery to one year after surgery
  Presence of post-operative trichiasis defined as at least one trichiatic eyelash or evidence of recent epilation. Trichiatic eyelashes are eyelashes touching the globe with the eye in primary gaze. The outcome will be assessed at 3, 6, 9 and 12 months. If the eyelid has trichiasis at 2 weeks, but not at any future visit, the eyelid will not be considered to have rPTT.

SECONDARY OUTCOMES:
Number of eyelids with moderate/severe eyelid contour abnormalities (ECA) | Assessed at last study visit (max: 2 years)
  The grader will assess for eyelid contour abnormalities (ECA) and grade the abnormalities as mild, moderate, or severe. For the analysis, no abnormality and mild eyelid contour abnormality will be combined, and moderate and severe eyelid contour abnormality will be combined. Results will be based on photograph grades.
  Category definitions are: 1) Mild: Vertical deviation from the natural contour, 1 mm in height (less than half the pupil height in daylight) and affecting 1/3 of horizontal eyelid length. 2) Moderate: Vertical deviation from the natural contour 1-2 mm in height (about the pupil height in daylight) or affecting 1/3-2/3 of horizontal eyelid length 3) Severe: Vertical deviation from the natural contour 2 mm in height (more than the pupil height in daylight) or a defect >2/3 of the horizontal eyelid length
Number of eyelids with clinically significant rPTT by twelve months | >2 weeks and up to 12 months after surgery
  Presence of clinically significant rPTT is defined as evidence of entropion AND either 1) >2 lashes touching the eye peripherally (Not touching the cornea in primary gaze) or 2) at least one eyelash emanating from the central portion of the eyelid, touching the cornea in primary gaze. Trichiatic eyelashes are eyelashes touching the globe with the eye in primary gaze. The outcome will be assessed at 3, 6, 9 and 12 months. If the eyelid has trichiasis at 2 weeks, but not at any future visit, the eyelid will not be considered to have rPTT.
Number of eyelids with rPTT by 24 months | Between two weeks and twenty four months after surgery
  Presence of repeat post-operative trichiasis defined as at least one trichiatic eyelash or evidence of recent epilation. Trichiatic eyelashes are eyelashes touching the globe with the eye in primary gaze. The outcome will be assessed at 3, 6, 9, 12, 18 and 24 months. If the eyelid has trichiasis at 2 weeks, but not at any future visit, the eyelid will not be considered to have rPTT.
Number of eyelids with each level of rPTT Severity | At first visit where rPTT is detected (up to 2 years after surgery)
  Severity will be graded as mild, moderate, or severe based on the number of eyelashes touching the globe and the amount of eyelashes epilated.
  Trichiasis severity will be defined using the following categories:
  * i. Mild: 1-4 eyelashes touching globe and no epilation OR <1/3 eyelashes epilated and no eyelashes touching the globe
  * ii. Moderate: 5-9 eyelashes touching globe and no epilation OR 1-4 eyelashes touching globe and <1/3 eyelashes epilated
  * iii. Severe: 5-9 eyelashes touching globe and <1/3 eyelashes epilated OR 10+ eyelashes touching globe (regardless of epilation status) OR ≥1/3 eyelashes epilated (regardless of eyelashes touching globe)
Cumulative number of eyelids with pyogenic granuloma | Any time between surgery and 24 months after surgery
  Pyogenic granulomas occasionally develop after trichiasis surgery. It is thought that this is a response to a foreign material, such as a sutures or an incision edge. All granulomas will be noted regardless of size. The investigators will count granulomas observed at the 3, 6, 9, 12, 18 and 24 month visit s(including participants where the granuloma was removed)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Gower, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- University of North Carolina, Chapel Hill, North Carolina, United States
- Kongwa Trachoma Project, Mtwara, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available at the time of publication of the primary and pre-planned secondary results papers.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual data that support the results will be shared beginning 9 and continuing for 36 months following publication.
Access Criteria: An investigator who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Kello AB, Merbs SL, Resnikoff S, West S, Mariotti SP, Solomon A. Trichiasis Surgery for Trachoma. 3rd ed. World Health Organization; 2024:80.
- [Background] Habtamu E, Wondie T, Aweke S, Tadesse Z, Zerihun M, Gashaw B, Roberts CH, Kello AB, Mabey DCW, Rajak SN, Callahan EK, Macleod D, Weiss HA, Burton MJ. Oral doxycycline for the prevention of postoperative trachomatous trichiasis in Ethiopia: a randomised, double-blind, placebo-controlled trial. Lancet Glob Health. 2018 May;6(5):e579-e592. doi: 10.1016/S2214-109X(18)30111-6. PMID 29653629
- [Background] Habtamu E, Wondie T, Aweke S, Tadesse Z, Zerihun M, Zewudie Z, Kello AB, Roberts CH, Emerson PM, Bailey RL, Mabey DC, Rajak SN, Callahan K, Weiss HA, Burton MJ. Posterior lamellar versus bilamellar tarsal rotation surgery for trachomatous trichiasis in Ethiopia: a randomised controlled trial. Lancet Glob Health. 2016 Mar;4(3):e175-84. doi: 10.1016/S2214-109X(15)00299-5. Epub 2016 Jan 14. PMID 26774708
- [Background] Burton MJ, Kinteh F, Jallow O, Sillah A, Bah M, Faye M, Aryee EA, Ikumapayi UN, Alexander ND, Adegbola RA, Faal H, Mabey DC, Foster A, Johnson GJ, Bailey RL. A randomised controlled trial of azithromycin following surgery for trachomatous trichiasis in the Gambia. Br J Ophthalmol. 2005 Oct;89(10):1282-8. doi: 10.1136/bjo.2004.062489. PMID 16170117
- [Background] Rajak SN, Habtamu E, Weiss HA, Kello AB, Gebre T, Genet A, Bailey RL, Mabey DC, Khaw PT, Gilbert CE, Emerson PM, Burton MJ. Absorbable versus silk sutures for surgical treatment of trachomatous trichiasis in Ethiopia: a randomised controlled trial. PLoS Med. 2011 Dec;8(12):e1001137. doi: 10.1371/journal.pmed.1001137. Epub 2011 Dec 13. PMID 22180732
- [Background] West SK, West ES, Alemayehu W, Melese M, Munoz B, Imeru A, Worku A, Gaydos C, Meinert CL, Quinn T. Single-dose azithromycin prevents trichiasis recurrence following surgery: randomized trial in Ethiopia. Arch Ophthalmol. 2006 Mar;124(3):309-14. doi: 10.1001/archopht.124.3.309. PMID 16534049
- [Background] Gower EW, West SK, Harding JC, Cassard SD, Munoz BE, Othman MS, Kello AB, Merbs SL. Trachomatous trichiasis clamp vs standard bilamellar tarsal rotation instrumentation for trichiasis surgery: results of a randomized clinical trial. JAMA Ophthalmol. 2013 Mar;131(3):294-301. doi: 10.1001/jamaophthalmol.2013.910. PMID 23494035
- [Background] Khandekar R, Mohammed AJ, Courtright P. Recurrence of trichiasis: a long-term follow-up study in the Sultanate of Oman. Ophthalmic Epidemiol. 2001 Jul;8(2-3):155-61. doi: 10.1076/opep.8.2.155.4165. PMID 11471085
- [Background] Khandekar R, Thanh TT, Luong VQ. The determinants of trichiasis recurrence differ at one and two years following lid surgery in Vietnam: A community-based intervention study. Oman J Ophthalmol. 2009 Sep;2(3):119-25. doi: 10.4103/0974-620X.57311. PMID 20927208
- [Background] Gower EW, Sisay A, Bayissasse B, Seyum D, Weaver J, Munoz B, Keil AP, Bankoski A, Sullivan KM, Kana H, Admassu F, Tadesse D, Merbs SL. The impact of modified incision height and surgical procedure on trichiasis surgery outcomes: Results of the maximizing trichiasis surgery success (MTSS) randomized trial. PLoS Negl Trop Dis. 2024 Sep 3;18(9):e0012034. doi: 10.1371/journal.pntd.0012034. eCollection 2024 Sep. PMID 39226693
- [Background] Courtright P, Gower EW, Kello AB, Solomon AW. Second Global Scientific Meeting on Trachomatous Trichiasis, Cape Town 4-6 November 2015. (Solomon A, ed.). World Health Organization; 2016.
- [Background] Merbs SL, Talero SL, Tadesse D, Sisay A, Bayissasse B, Weaver JU, Gower EW. A New Surgical Technique for Postoperative Trachomatous Trichiasis. Ophthalmic Plast Reconstr Surg. 2021 Nov-Dec 01;37(6):595-598. doi: 10.1097/IOP.0000000000002055. PMID 34570049
- [Background] Gower EW, West SK, Cassard SD, Munoz BE, Harding JC, Merbs SL. Definitions and standardization of a new grading scheme for eyelid contour abnormalities after trichiasis surgery. PLoS Negl Trop Dis. 2012;6(6):e1713. doi: 10.1371/journal.pntd.0001713. Epub 2012 Jun 26. PMID 22745845
- [Background] Kamuyu MK, Kelly M, Somerville S. A secondary analysis to determine countries and districts eligible for documented full geographic coverage for trichiasis case finding and outreaches. Int Health. 2023 Dec 4;15(15 Suppl 2):ii53-ii57. doi: 10.1093/inthealth/ihad075. PMID 38048374